CLINICAL TRIAL: NCT07389941
Title: Semaglutide PrIor to CathEeter Ablation in Patients With Atrial Fibrillation (SPICE-AF)
Brief Title: Semaglutide PrIor to CathEeter Ablation in Patients With Atrial Fibrillation
Acronym: SPICE-AF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Roland Richard Tilz, MD, Director, Department of Rhythmology, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPICE_AF
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation | interventions — semaglutide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Catheter ablation for atrial fibrillation plus semaglutide (Experimental): Catheter ablation for atrial fibrillation plus semaglutide (up to 2.4 mg weekly)
  Interventions: Drug: Semaglutide (SEMA)
- Catheter ablation for atrial fibrillation and no glucacon-like peptide-1 receptor therapy (No Intervention): Catheter ablation for atrial fibrillation and no glucacon-like peptide-1 receptor therapy (standard therapy)

INTERVENTIONS:
Drug: Semaglutide (SEMA) — Catheter ablation for AF plus semaglutide (up to 2.4 mg weekly)
  Arms: Catheter ablation for atrial fibrillation plus semaglutide

SUMMARY:
To evaluate whether pre-treatment with semaglutide is superior to standard care in improving freedom from atrial fibrillation (AF) at 12 months following catheter ablation in patients with obesity and symptomatic AF undergoing first-time ablation.

ELIGIBILITY:
Inclusion criteria:

* Age 18-80 years
* Symptomatic paroxysmal or persistent AF eligible for first-time catheter ablation
* Body mass index ≥30 kg/m or body mass index ≥28 kg/m plus ≥1 weight-related comorbidity
* No prior treatment with glucacon-like peptide-1 receptor agonists

Exclusion criteria:

* Current use of glucacon-like peptide-1 receptor agonists or dipeptidyl peptidase 4 inhibitors or use within the last 90 days prior to screening
* Current antiobesity medication use or use within the last 90 days prior to screening
* A self-reported change in body weight of >5 kg within 30 days before screening
* History of bariatric surgery
* History of diabetes mellitus
* Hospitalization for unstable angina, or transient ischemic attack <30 days prior to screening
* Pulmonary embolism <90 days before screening
* Myocardial infarction, or stroke <90 days prior to screening
* Uncontrolled thyroid disease: thyroid-stimulating hormone >10.0 mIU/L or <0.4 mIU/L at screening
* Active malignancy
* Acute pancreatitis <180 days before screening
* History or presence of chronic pancreatitis
* Chronic kidney disease with creatinine clearance <30 mL/min
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* Chronic inflammatory conditions requiring immunosuppression and/or on glucocorticoids
* Pregnancy, breast-feeding or planning pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmia (AF/atrial flutter/atrial tachycardia >30 sec) at 12 months post-ablation (8-week-blanking period) | 12 months

IPD SHARING:
Plan to Share IPD: No